CLINICAL TRIAL: NCT06247696
Title: Sweet Scents to Sweet Dreams: Use of Herbal Pillows to Facilitate Sleep and Improve Quality of Life
Brief Title: Sweet Scents to Sweet Dreams
Acronym: SSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: Cura Rest/Healing and Yoga Arts (Unknown)
Responsible Party: Principal Investigator, Paula Witt-Enderby, Professor of Pharmacology, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023/11/25
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disturbance; Mental Health Issue
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo Pillow (Placebo Comparator)
  Interventions: Other: Herbal Pillows
- Control Pillow (Active Comparator)
  Interventions: Other: Herbal Pillows
- Vata Pillow (Experimental)
  Interventions: Other: Herbal Pillows
- Pitta Pillow (Experimental)
  Interventions: Other: Herbal Pillows
- Kapha Pillow (Experimental)
  Interventions: Other: Herbal Pillows

INTERVENTIONS:
Other: Herbal Pillows — Pillows containing herbs

SUMMARY:
The purpose of this study is to determine the effect of herbal pillows on sleep and quality of life in a healthy population using actigraphy, validated questionnaires and daily diary logs. The goal of this study is to improve sleep and quality of life using herbal and Ayurveda/holistic-based botanical pillows.

ELIGIBILITY:
Inclusion Criteria:

* You must be at least 18 years of age.
* You must be willing to adhere to a sleep hygiene protocol (e.g., 10pm-midnight-6-8am) for 2 weeks without interruption in the comfort of your home.
* You must be willing to wear a watch that monitors your sleep and light as well as a sleep mask for two consecutive weeks.
* During the testing period, you must be willing to refrain from alcohol and anything that can affect mood and sleep.
* You must allow for the placement of an herbal pillow next to your head while sleeping for one week during testing.
* You must be willing to fill out short sleep logs during the 2 weeks of testing.
* You must also be willing to come to the study location on 3 occasions over a 2 week period.

Exclusion Criteria:

* Males or females with any condition that prevents adequate inhalation of botanical pillows [e.g., Chronic Obstructive Pulmonary Disease (COPD), use of a Continuous Positive Airway Pressure (CPAP), deviated septum, etc].
* Males or females on mood altering substances prescription (e.g., anti-depressants, anxiolytics, Ritalin, Adderall, anti-convulsants; opioids, etc), non-prescription/over-the-counter (OTC) drugs/herbal/natural products [(e.g., tetrahydrocannabinol (THC)-containing compounds, melatonin, St. John's Wort, lavender capsules, essential oils, perfume-containing products, etc].
* Any environmental, physical condition or pathology that can significantly impact on sleep and prevent an approximate 10pm-midnight-6-8am sleep rhythm (e.g., shift work, studying/exams, rotations, insomnia, new parents, nocturia, restless leg syndrome, chronic pain, etc).
* Any medications that can influence sleep [(e.g., use of beta blockers; anti-histamines; dexamethasone; angiotensin converting enzyme inhibitor (ACEI); nicotine products, alpha blockers]
* Chemical sensitivities
* Allergies
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Function | 2 weeks
  Assessments of rest/activity rhythms by wrist actigraphy

SECONDARY OUTCOMES:
Subject-reported effects on sleep | 2 weeks
  Assessments will be made using the validated sleep questionnaire, Pittsburgh Sleep Quality Index, PSQI
Subject-reported effects on depression | 2 weeks
  Assessments will be made using the validated depression questionnaire, Center for Epidemiology Studies-Depression, CES-D
Subject-reported effects on anxiety | 2 weeks
  Assessments will be made using the validated anxiety questionnaire, Spielberg State-Trait Anxiety Inventory, STAI
Subject-reported effects on stress | 2 weeks
  Assessments will be made using the validated stress questionnaire, Perceived Stress Scale, PSS
Subject-reported effects on quality of life | 2 weeks
  Assessments will be made using the validated health-related quality of life questionnaire, quality of life (Health-related Quality of Life, HR-QOL
Ayurvedic assessments of doshas | 2 weeks
  Assessment of dosha-specific herbal pillows on dosha balancing

CONTACTS AND LOCATIONS:
Overall Officials: Paula A. Witt-Enderby, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request